CLINICAL TRIAL: NCT02588196
Title: The Relationships Between Gene Polymorphisms of LTA4H and Dexamethasone Treatment for Tuberculous Meningitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hui Bu (Other)
Responsible Party: Sponsor-Investigator, Hui Bu, chief physician, Hebei Medical University
Organization: Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH 002
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Tuberculous Meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — dexamethasone acetate

ARMS (1):
- treatment of dexamethasone group (Experimental)
  Interventions: Drug: Dexamethasone acetate

INTERVENTIONS:
Drug: Dexamethasone acetate

SUMMARY:
The study aimed to evaluate the relationships between the gene polymorphisms of leukotriene A4 hydrolase(LTA4H) and Dexamethasone treatment for tuberculous meningitis in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

patients were eligible to enter the study if they met the diagnositic criteria for possible, probable or definite Tuberculosis meningitis(TBM).

Exclusion Criteria:

Patients were excluded if they were infected with HIV, diagnosed as carcinomatous meningitis, viral meningitis, purulent meningitis, cryptococcus meningitis.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
MRI | 6 month
  whether MRI show infarction, hydrocephalus, meningeal enhancement
changes of cerebrospinal fluid | 1 year
changes of clinical symptoms | 1 year
  headache duration, duration of fever,presence of cranial nerve damage